CLINICAL TRIAL: NCT06152718
Title: New Regenerative and Anti-aging Medicine Approach Based on Single Strand Alpha-1 Collagen for Neo-collagenesis Induction: Clinical and Instrumental Experience of a New Medical Device for Dermal Regeneration (Karisma)
Brief Title: New Regenerative Approach for Dermal Renovation (Karisma)
Acronym: Karisma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Novi Sad, Faculty of Sport and Physical Education (Other); Patrizia Proia, University of Palermo (Unknown); Filippo Castrogiovanni, Taumedika s.r.l (Unknown); Antonino De Pasquale, University of Catania (Unknown); Luigi Di Rosa, University of Palermo (Unknown); Sara Baldassano, University of Palermo (Unknown)
Responsible Party: Principal Investigator, Sonya Vasto, Associate professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49-10-02-2023-1
Record Dates: First submitted 2023-11-07; First posted 2023-12-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2023-12

CONDITIONS: Skin Manifestations
Keywords: regenerative medicine; skin ageing; collagen production; filler; Hyaluronic acid; inflammation
MeSH Terms: conditions — Skin Manifestations; Inflammation

STUDY DESIGN:
Intervention Model Description: the group of researchers will assess partecipants before the intervention (baseline measurement) and then again after the intervention. The change from baseline to the end of the study can be attributed to the intervention.There is no separate control group for comparison.
Masking Description: single-group study cannot blind the occurred intervention: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Karisma arm (Experimental): Selected participant (inclusion criteria) undergo one injection of single-strand alpha 1 collagen (3ml)
  Interventions: Other: Karisma

INTERVENTIONS:
Other: Karisma — Use of regenerative capabilities of a new medical device focused on dermal redensification, induced by injections of single-strand alpha 1 collagen

SUMMARY:
Purpose/Objectives of the Study: Regenerative medicine, as well as aesthetic plastic surgery and dermatology field persistently seeks innovative, minimally invasive interventions to enhance skin quality and mitigate signs of aging. This study evaluates the regenerative capabilities of a new medical device focused on dermal redensification, induced by injections of single-strand alpha 1 collagen, to verify its ability, in a specific formulation (contained within a matrix of hyaluronic acid and carboxymethylcellulose), to induce dermal stimulation in both scar outcomes and regenerative medicine applied to skin aging.

DETAILED DESCRIPTION:
Study Population (including any inclusion/exclusion criteria): : A total of 100 patients, aged between 25 and 70 years of both sexes, subdivided into 3 demographically similar subgroups, will be assessed in this exploratory study. The intervention entailed the administration of the single-strand alpha 1 collagen - hyaluronic acid soft filler, with subsequent evaluations employing the Antera 3D® skin scanner and two multiple choice questionnaires, FACE-Q and Global Aesthetic Improvement Scale (GAIS) to obtain objective data and subjective evaluations recorded by patients. All patients must be in good general health. not affected by oncological, rheumatological, chronic inflammatory diseases (including dermatitis, psoriasis, etc.). patients should not take systemic drugs during the course of the aforementioned study. The sample size of 100 patients is in line with studies already carried out in this field, in order to obtain adequate statistical power, also in anticipation of a physiological drop out of some patients. Parametric and non-parametric tests will be used to test the results to assess the significance of discrete and continuous numerical variables, as well as descriptive statistics for all patient groups.

Within the scope of this project, the investigators plan to recruit four cohorts of subjects:

1. smokers (30 subjects)
2. non-smokers (30 subjects)
3. subjects affected by acne scars (40)

All patients must be in general good health, not affected by oncological, rheumatological, allergic, chronic inflammatory diseases (including dermatitis, psoriasis, etc.). Patients should not have metabolic or cardiovascular diseases, should not have received other injections of hyaluronic acid or similar substances for at least 6 months before the start of treatment, and should not take systemic drugs during the study.

The primary endpoints will be those to evaluate the subjective changes in texture, hydration, compactness, brightness, and quality of skin roughness through the administration of multiple-choice tests already validated by numerous scientific studies (Global Aesthetic Improvement Scale GAIS; FACE-Q Age Appearance Appraisal) and objective changes through non-invasive measurements, such as dermal thickness by high-frequency ultrasound; the depth of wrinkles, amount of melanin and hemoglobin through 3D Antera Scanner, to assess the regenerative capabilities of the medical device in patients affected by acne scars, in the atrophic and dystrophic skin alterations of the body, as well as in the photo and chronoaging of the skin of the face, neck, and décolleté in smoking and non-smoking patients.

As a secondary endpoint, it will be analyzed through a Raman spectroscope whether the changes induced by the product will be able to modify the local skin oxidative-reductive picture through spectroscopic analysis on the skin of dermal carotenoids. Furthermore, tissue biopsy will be colected in order to analyze changes in tissue structure, including collagen deposition and stromal characteristics.

Study Procedures: Participants will undergo the following tests :

t0: instrumental evaluation, initial parameter recording, administration of clinical evaluation tests, photographic iconography, biopsies and first injection of Karisma.

t1: first check after 15 days, instrumental evaluation, administration of clinical evaluation tests, photographic iconography.

t2: second check 30 days after the first injection of Karisma, instrumental evaluation, administration of clinical evaluation tests, photographic iconography, second injection of Karisma.

t3: third check 60 days after the first injection of Karisma, instrumental evaluation, administration of clinical evaluation tests, photographic iconography and biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-65 years old
* skin ageing evidences from mild to severe

Inclusion Criteria:

* not affected by oncological diseases
* rheumatological diseases
* no allergic diseases
* no chronic inflammatory diseases (including dermatitis, psoriasis, etc.). Patients should not have;
* metabolic diseases
* cardiovascular diseases,
* should not have received other injections of hyaluronic acid or similar substances for at least 6 months before the start of treatment,
* should not take systemic drugs during the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
"Change from Baseline to day 15 in the mean depth of skin wrinkles (mm) | baseline and day 15
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar, in a portion of skin selected by the investigator. skin depth is expressed in millimeters.
"Change from Baseline to day 30 in the mean depth of skin wrinkles (mm) | baseline and day 30
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar, in a portion of skin selected by the investigator. skin depth is expressed in millimeters.
"Change from Baseline to day 60 in the mean depth of skin wrinkles (mm) | baseline and day 60
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar, in a portion of skin selected by the investigator. skin depth is expressed in millimeters.
"Change from Baseline to day 15 in melanin quantity ( arbitrary unit from 0.1-1 indicated by Antera 3D scanner) | baseline and day 15
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar; Melanin values are expressed in arbitrary values ranging from 0.1 to 1
"Change from Baseline to day 30 in melanin quantity ( arbitrary unit from 0.1-1 indicated by Antera 3D scanner) | baseline and day 30
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar; Melanin values are expressed in arbitrary values ranging from 0.1 to 1
"Change from Baseline to day 60 in melanin quantity ( arbitrary unit from 0.1-1 indicated by Antera 3D scanner) | baseline and day 60
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure depth of skin lines, wrinkles and acne scar; Melanin values are expressed in arbitrary values ranging from 0.1 to 1
"Change from Baseline to day 15 in hemoglobin quantity. | baseline and day 15
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure hemoglobin values that are expressed in arbitrary values ranging from 0.1 to 4
"Change from Baseline to day 30 in hemoglobin quantity. | baseline and day 30
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure hemoglobin values that are expressed in arbitrary values ranging from 0.1 to 4
"Change from Baseline to day 60 in hemoglobin quantity. | baseline and day 60
  changes will be evaluated using 3D Antera Scanner. It is a validated skin device that is used to measure hemoglobin values that are expressed in arbitrary values ranging from 0.1 to 4
"Change from Baseline in the Mean values of FACE-Q questionnaire at 15 days" | baseline and day 15
  FACE-Q questionnaire is a validated multiple choices questionnaire used to assess patient aging appraisaland perceived skin quality of face and neck. Test will be provided to patients at baseline and after 15 days in order to evaluate if any perceived changes are present. 47 questions will be provided. Every question has a 4 values answer ranging from 1 (I.E. very dissatisfied) to 4 (I.E. very satisfied).
"Change from Baseline in the Mean values of FACE-Q questionnaire, at 30 days" | baseline and day 30
  FACE-Q questionnaire is a validated multiple choices questionnaire used to assess patient aging appraisaland perceived skin quality of face and neck. Test will be provided to patients at baseline and after 15 days in order to evaluate if any perceived changes are present. 47 questions will be provided. Every question has a 4 values answer ranging from 1 (I.E. very dissatisfied) to 4 (I.E. very satisfied).
"Change from Baseline in the Mean values of FACE-Q questionnaire, at 60 days" | baseline and day 60
  FACE-Q questionnaire is a validated multiple choices questionnaire used to assess patient aging appraisaland perceived skin quality of face and neck. Test will be provided to patients at baseline and after 15 days in order to evaluate if any perceived changes are present. 47 questions will be provided. Every question has a 4 values answer ranging from 1 (I.E. very dissatisfied) to 4 (I.E. very satisfied).
"Change from Baseline in the Mean values of GAIS Global Aesthetic Improvment Scale, at 15 days" | baseline and day 15
  The GAIS Global Aesthetic Improvement Scale, is a validated five-point scale for assessing global aesthetic improvement in appearence compared to pretratment. The ratings range from "very much improved", "much improved" "improved", unchanged and worsened.
"Change from Baseline in the Mean values of GAIS Global Aesthetic Improvment Scale, at 30 days" | baseline and day 30
  The GAIS Global Aesthetic Improvement Scale, is a validated five-point scale for assessing global aesthetic improvement in appearence compared to pretratment. The ratings range from "very much improved", "much improved" "improved", unchanged and worsened.
"Change from Baseline in the Mean values of GAIS Global Aesthetic Improvment Scale, at 60 days" | baseline and day 60
  The GAIS Global Aesthetic Improvement Scale, is a validated five-point scale for assessing global aesthetic improvement in appearence compared to pretratment. The ratings range from "very much improved", "much improved" "improved", unchanged and worsened.

SECONDARY OUTCOMES:
tissue Biopsies | baseline and day 60
  Core needle biopsies to evaluate histological changes in ageing tissues

CONTACTS AND LOCATIONS:
Locations (2):
- NabBio, Palermo, PA, Italy
- University of Novi Sad, Serbia, Novi Sad, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad S, Galadari H, Patil A, Goldust M, Al Salam S, Guida S. Evaluation of the biostimulatory effects and the level of neocollagenesis of dermal fillers: a review. Int J Dermatol. 2022 Oct;61(10):1284-1288. doi: 10.1111/ijd.16229. Epub 2022 Apr 29. PMID 35486036
- [Background] Fallacara A, Manfredini S, Durini E, Vertuani S. Erratum: Hyaluronic Acid Fillers in Soft Tissue Regeneration. Facial Plast Surg. 2017 Apr;33(2):244. doi: 10.1055/s-0037-1601851. Epub 2017 Apr 7. No abstract available. PMID 28388806
- [Background] Kapoor KM, Saputra DI, Porter CE, Colucci L, Stone C, Brenninkmeijer EEA, Sloane J, Sayed K, Winaya KK, Bertossi D. Treating Aging Changes of Facial Anatomical Layers with Hyaluronic Acid Fillers. Clin Cosmet Investig Dermatol. 2021 Aug 26;14:1105-1118. doi: 10.2147/CCID.S294812. eCollection 2021. PMID 34471372
- [Background] Bukhari SNA, Roswandi NL, Waqas M, Habib H, Hussain F, Khan S, Sohail M, Ramli NA, Thu HE, Hussain Z. Hyaluronic acid, a promising skin rejuvenating biomedicine: A review of recent updates and pre-clinical and clinical investigations on cosmetic and nutricosmetic effects. Int J Biol Macromol. 2018 Dec;120(Pt B):1682-1695. doi: 10.1016/j.ijbiomac.2018.09.188. Epub 2018 Oct 1. PMID 30287361
- [Background] Vasvani S, Kulkarni P, Rawtani D. Hyaluronic acid: A review on its biology, aspects of drug delivery, route of administrations and a special emphasis on its approved marketed products and recent clinical studies. Int J Biol Macromol. 2020 May 15;151:1012-1029. doi: 10.1016/j.ijbiomac.2019.11.066. Epub 2019 Nov 9. PMID 31715233
- [Background] Iaconisi GN, Lunetti P, Gallo N, Cappello AR, Fiermonte G, Dolce V, Capobianco L. Hyaluronic Acid: A Powerful Biomolecule with Wide-Ranging Applications-A Comprehensive Review. Int J Mol Sci. 2023 Jun 18;24(12):10296. doi: 10.3390/ijms241210296. PMID 37373443
- [Background] Ricard-Blum S. The collagen family. Cold Spring Harb Perspect Biol. 2011 Jan 1;3(1):a004978. doi: 10.1101/cshperspect.a004978. PMID 21421911
- [Background] Avila Rodriguez MI, Rodriguez Barroso LG, Sanchez ML. Collagen: A review on its sources and potential cosmetic applications. J Cosmet Dermatol. 2018 Feb;17(1):20-26. doi: 10.1111/jocd.12450. Epub 2017 Nov 16. PMID 29144022
- [Background] Chattopadhyay S, Raines RT. Review collagen-based biomaterials for wound healing. Biopolymers. 2014 Aug;101(8):821-33. doi: 10.1002/bip.22486. PMID 24633807
- [Background] Rapaport MJ, Salit R, Rivkin L. Collagen injections for aging skin lines (wrinkles). J Am Acad Dermatol. 1984 Aug;11(2 Pt 1):250-2. doi: 10.1016/s0190-9622(84)70159-9. PMID 6480926
- [Background] Lucey P, Goldberg DJ. Complications of collagen fillers. Facial Plast Surg. 2014 Dec;30(6):615-22. doi: 10.1055/s-0034-1396904. Epub 2014 Dec 23. PMID 25536127
- [Background] Cui Y, Wang F, Voorhees JJ, Fisher GJ. Rejuvenation of Aged Human Skin by Injection of Cross-linked Hyaluronic Acid. Plast Reconstr Surg. 2021 Jan 1;147(1S-2):43S-49S. doi: 10.1097/PRS.0000000000007620. PMID 33347074
- [Background] Wells JM, Gaggar A, Blalock JE. MMP generated matrikines. Matrix Biol. 2015 May-Jul;44-46:122-9. doi: 10.1016/j.matbio.2015.01.016. Epub 2015 Jan 28. PMID 25636538
- [Background] Maquart FX, Bellon G, Pasco S, Monboisse JC. Matrikines in the regulation of extracellular matrix degradation. Biochimie. 2005 Mar-Apr;87(3-4):353-60. doi: 10.1016/j.biochi.2004.10.006. PMID 15781322
- [Background] Wu GT, Kam J, Bloom JD. Hyaluronic Acid Basics and Rheology. Facial Plast Surg Clin North Am. 2022 Aug;30(3):301-308. doi: 10.1016/j.fsc.2022.03.004. PMID 35934432